CLINICAL TRIAL: NCT02917954
Title: Full Evaluation, Scale and Spread: Pragmatic Trial of the HSPRN-Bridgepoint Electronic Patient Reported Outcome (ePRO) Mobile Application to Support the Needs of Persons With Complex Chronic Disease and Disability
Brief Title: Electronic Patient Reported Outcome (ePRO) Mobile Application Pragmatic Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: University of Toronto (Other); Ottawa Hospital Research Institute (Other); QoC Health Inc. (Unknown)
Responsible Party: Principal Investigator, Carolyn Steele Gray, Post-doctoral Fellow, Scientific Lead, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ePRO2016
Record Dates: First submitted 2016-09-13; First posted 2016-09-28 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Chronic Disease; Quality of Life
Keywords: eHealth/mHealth solutions; complex care needs; seniors; patient-centred care; goal-oriented care; primary health care; implementation; pragmatic trial; health outcomes; cost-effectiveness analysis
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Stepped-wedge randomized trial. Group 1: 3 month control period followed by a 12 month intervention period. Group 2: 6 month control period followed by a 9 month intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ePRO Control (3 or 6 months) (No Intervention): Control participants will complete surveys at baseline, 3 months, and/or 6 months. Surveys will capture patient demographics, their assessment of quality-of-life, chronic disease management, and primary care experience. A part from completing these surveys, no change to routine care will be seen.
- ePRO intervention (12 or 9 months) (Experimental): During the ePRO Tool intervention participants will complete surveys at every 3 months intervals starting month at 4 or month 7, for study duration. Surveys capture patient demographics, assessment of quality-of-life, chronic disease management, primary care experience, and Electronic Patient Reported Outcome (ePRO) Mobile Application tool usability.
  Participants will also meet with their provider to setup and monitor a health goal to track during the study via the ePRO application. During the study, participants will meet with their primary care providers 4-5 times to discuss their health goal monitoring. Post-study participants will discuss their experience using the ePRO app in an interview or focus group setting.
  Interventions: Device: ePRO Tool Intervention

INTERVENTIONS:
Device: ePRO Tool Intervention — The ePRO tool includes two features: 1) My Goal Tracker and 2) Health Journal. My Goal Tracker allows patients and providers to collaboratively create goal-oriented patient care-plans, and helps patients to track outcomes related to their goals using a mobile device. The Health Journal allows patients, their caregivers and primary care providers to monitor patients' symptoms and outcomes.
  Other Names: Electronic Patient Reported Outcome Mobile Application; ePRO
  Arms: ePRO intervention (12 or 9 months)

SUMMARY:
Canadian and international health care systems require solutions on how to address the needs of a relatively small population that take up a large portion of health care resources. In Ontario, 10% of the population accounts for 79% of total system costs, with similar trends found in other parts of Canada and internationally. Most high-cost users are seniors, older adults, with multiple chronic conditions and complex care needs who are living in the community. Beyond the cost issues, older adults experiencing multi-morbidity are at higher-risk of poor health outcomes and experience lower quality of life as compared to individuals experiencing single illness only.

Since April 2013 the electronic Patient Reported Outcomes (ePRO) mobile application and portal, has undergone a multi-phased, user-centred design evaluation approach to develop a tool designed to meet the needs of older adults with complex care needs and their primary care providers. The ePRO tool is designed to collect person-centred, person-reported indicators to improve care by supporting primary care delivery and enhancing patient self-management.

The ePRO tool includes two features: 1) My Goal Tracker and 2) Health Journal. My Goal Tracker allows patients and providers to collaboratively create goal-oriented patient care-plans, and helps patients to track outcomes related to their goals using a mobile device. The Health Journal allows patients, their caregivers and primary care providers to monitor patients' symptoms and outcomes. The ePRO tool was re-evaluated and modified following each previous study phase (I-IV). This project marks the final phase of the study in which the investigators will conduct a pragmatic trial of the ePRO tool in 8-16 Family Health Teams in Ontario through a stepped-wedge randomized trial with an embedded case study. In this evaluation of the tool the investigators will assess outcome, process and context measures to identify how the tool affects patients, providers and the system at point-of-care.

DETAILED DESCRIPTION:
The pragmatic trial will take place at 6 Family Health Teams (FHTs) to a maximum of 16 FHTs in Ontario utilizing a stepped-wedge randomized method with an embedded case study of implementation at four sites. The research team will observe provider-patient goal-setting visits at the time of onboarding onto the intervention. Additional consent will be obtained from the patient and provider prior to initiating the observational visit. In addition, the research team will attend FHT rounds at the identified case study sites (when appropriate) to observe and document how providers discuss and set goals in an interdisciplinary team environment. Using a stepped-wedge design, each FHT will receive the ePRO tool (intervention) but will be randomized on when in the stepped-wedge design they will receive the intervention. The stepped-wedge randomization will assign (through number generator or coin flip) each of the FHTs to either a: 1) 3 month control period and a 12 month intervention period, or 2) 6 month control period and a 9 month intervention period; and their respective participants will be assigned accordingly.

Providers and patients recruited at all sites will receive training on how to use the ePRO tool prior to the start of the trial. During the intervention period, patients will receive one-on-one training with a research assistant; and provider training will occur in a group setting. Training will be led by a member of the research team and will take between 30-60 minutes. Patients and providers will also be provided with a manual and training video on how to use the tool and portal, and the patients will be offered refresher sessions (individual or group) every 3 months over the duration of the study.

Following consent, all patients will complete pre and post surveys every 3 months (through control and intervention periods). Patients will also complete an additional survey at study closeout to capture tool usability feedback. We anticipate survey completion to take 20-35 minutes.

Additionally, patients are requested to attend a minimum of two schedule appointments with their provider during the study. The first (on-boarding) visit will have the patient and provider collaboratively discuss and set monitoring protocols for tracking. The second (off-boarding) visit, following the monitoring period, will allow patients and providers to privately discuss their experience with the ePRO tool, before participating in their respective focus group or interview. As was the case in our usability pilot and exploratory trial, we anticipate that patients will have additional appointments with their providers during the study at which point they can use the tool to discuss patient progress towards goals. All patients are requested to attend 4-5 scheduled appointments with their provider during the study. In accordance to earlier study phases on-boarding and off-boarding visits typically take 30 minutes. Other scheduled visits take between 10-30 minutes depending on the type of visit and provider they are seeing.

Embedded within the pragmatic trial will be case studies of 4 intervention sites. Provider and patient participants at case sites will participate in mid and post-intervention period semi-structured interviews to capture implementation enables and barriers. To adequately capture organizational level barriers and enablers we will additionally conduct semi-structured interviews with organizational leaders (executive directors and/or clinical leads). We will also collect relevant documents from all sites (i.e. organizational policies regarding the use of mobile applications or provider trainings and manuals in using technology as part of usual care).

This described stepped-wedge design is an update from the initially conceived pragmatic cluster trial of 22 sites. This shift was necessary due to site recruitment challenges experienced, in particular that sites did not want to be recruited to the study unless they could use the technology. As such a stepped-wedge trial was deemed more appropriate. With this new design the updated power calculation for the study indicated a new target of 176 patients across sites whereas the initial calculation was for 660.

Stepped-wedge sample size calculation:

Minimum sample size required for the recruitment of sites and patients was determined using closed-form analytical formulae with a power of 80% based on: a minimal clinically important difference of our core measure of quality of life (the AQoL-4D) of 0.06, an expected standard deviation in AQoL of 0.22, an expected ICC of 0.01 (calculated based on total primary care utilization over a one year period among a 10% sample of the Ontario population, which served here as a proxy measure for patient outcomes), and an expected attrition rate of 10% (rated based on previous studies in similar population groups using similar technology). A minimum sample size of 176 patients was calculated.

ELIGIBILITY:
Inclusion Criteria:

1. a FHT patient at one of the FHT sites selected and is 60 years or older;
2. physical capability to use a tablet and/or a caregiver who can use the tablet on their behalf;
3. ability to read and write in English and/or the availability of a caregiver who can do so on their behalf;
4. has complex care needs defined as two or more chronic conditions and 10 or more visits to their primary health care provider within the last 12 months; and
5. be thinking about or ready to make changes to support their self-management.

In addition patients can self-identify and join the study, as well as providers can identify other patients they feel fit our eligibility criteria that may not have been pulled from the EMR system. This allows eligible patients to enroll into the study that may have been missed when identifying patients through the EMR system.

Exclusion Criteria:

1. Absence of Inclusion Criteria

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline Assessment of Quality-of-Life at 3 month intervals for 15 months | Baseline, 3 months, 6 months, 9 months, 12 months, and study end (15-months)
  Our primary measure of patient oriented outcome is quality of life measured by the Assessment for Quality of Life Scale.
  12 Item survey, with each item having 4 response levels.

SECONDARY OUTCOMES:
ePRO cost-effectiveness - health system perspective | 15-months
  Only costs that are borne to the government, such as costs of intervention and costs of health services incurred during the 1-year follow-up period will be considered. Costs of the intervention will be estimated based on anticipated real-world licensing and ongoing costs for: software access, hosting and data management, program support and device management, application support, training, incremental data plan(s) (depending on volume of use in the intervention group), and for the Cloud Connect platform.
Patient Demographic and Characteristic information | Baseline
  We will capture patient demographic and characteristic information such as age, gender, ethnicity, chronic illness profile, socio-economic status, and IT skills using the Patient Demographic forms.
Provider Demographic and Characteristic Information | Baseline
  We will capture provider demographic and characteristic information such as age, gender, ethnicity, chronic illness profile, socio-economic status, and IT skills using the Provider Demographic forms.
Change from baseline Patient/Caregiver Self-Reported Costs at 3 month intervals for study duration (15 months) | Baseline, 3 months, 6 months, 9 months, 12 months, and study-end (15-months)
  Patient/Caregiver Self-Reported Costs form will provide contextual information about our users to support data analysis.
  Responses will be captured using a 6-point Likert scale.
Change from baseline Patient Experience at 3 month intervals for study duration (15 months) | Baseline, 3 months, 6 months, 9 months,12 months, and study-end (15-months)
  Patient Experience will be captured from the patient-experience survey distributed by the Family Health Teams of Ontario Association (AFHTO) to all Family Health Teams.
  3 Item survey, with responses captured on a 5-point Likert scale
Change from baseline Patient Activation Measure at 3 month intervals for study duration (15 months) | Baseline, 3 months, 6 months, 9 months, 12 months, and study-end (15-months)
  Patient Self-Management will be captured by the 13-Item Patient Activation Measure. Each item will have a 5-point Likert scale response level.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Steele Gray, PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Dr. Carolyn Steele Gray, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The reported data (which includes patient information at the aggregate level) will be disseminated widely via reports, conference presentations, peer reviewed journal articles and other standard modes of knowledge translation.
Supporting Information: CSR
Time Frame: Data will be available through open access journal publications anticipated in the year 2020
Access Criteria: Open access peer reviewed journal publication
URL: http://eproapp.weebly.com/

REFERENCES:
- [Background] Commission on the Reform of Ontario's Public Services, Public Services for Ontarians: A Path to Sustainability and Excellence. 2012.
- [Background] Reid R, Evans R, Barer M, Sheps S, Kerluke K, McGrail K, Hertzman C, Pagliccia N. Conspicuous consumption: characterizing high users of physician services in one Canadian province. J Health Serv Res Policy. 2003 Oct;8(4):215-24. doi: 10.1258/135581903322403281. PMID 14596756
- [Background] Heslop L, Athan D, Gardner B, Diers D, Poh BC. An analysis of high-cost users at an Australian public health service organization. Health Serv Manage Res. 2005 Nov;18(4):232-43. doi: 10.1258/095148405774518633. PMID 16259671
- [Background] Department of Health, Long Term Conditions Compedium of Information, Third Edition, D.o. Health, Editor. 2012: United Kingdom.
- [Background] Emanuel EJ. Where are the health care cost savings? JAMA. 2012 Jan 4;307(1):39-40. doi: 10.1001/jama.2011.1927. No abstract available. PMID 22215161
- [Background] Rosella LC, Fitzpatrick T, Wodchis WP, Calzavara A, Manson H, Goel V. High-cost health care users in Ontario, Canada: demographic, socio-economic, and health status characteristics. BMC Health Serv Res. 2014 Oct 31;14:532. doi: 10.1186/s12913-014-0532-2. PMID 25359294
- [Background] Marengoni A, Angleman S, Melis R, Mangialasche F, Karp A, Garmen A, Meinow B, Fratiglioni L. Aging with multimorbidity: a systematic review of the literature. Ageing Res Rev. 2011 Sep;10(4):430-9. doi: 10.1016/j.arr.2011.03.003. Epub 2011 Mar 23. PMID 21402176
- [Background] Bayliss EA, Bosworth HB, Noel PH, Wolff JL, Damush TM, Mciver L. Supporting self-management for patients with complex medical needs: recommendations of a working group. Chronic Illn. 2007 Jun;3(2):167-75. doi: 10.1177/1742395307081501. PMID 18083671
- [Derived] Tahsin F, Austin T, McKinstry B, Mercer SW, Loganathan M, Thavorn K, Upshur R, Steele Gray C. Examining Use Behavior of a Goal-Supporting mHealth App in Primary Care Among Patients With Multiple Chronic Conditions: Qualitative Descriptive Study. JMIR Hum Factors. 2022 Nov 30;9(4):e37684. doi: 10.2196/37684. PMID 36449335
- [Derived] Miranda RN, Bhuiya AR, Thraya Z, Hancock-Howard R, Chan BC, Steele Gray C, Wodchis WP, Thavorn K. An Electronic Patient-Reported Outcomes Tool for Older Adults With Complex Chronic Conditions: Cost-Utility Analysis. JMIR Aging. 2022 Apr 20;5(2):e35075. doi: 10.2196/35075. PMID 35442194
- [Derived] Singh H, Tahsin F, Nie JX, McKinstry B, Thavorn K, Upshur R, Harvey S, Wodchis WP, Gray CS. Exploring the perspectives of primary care providers on use of the electronic Patient Reported Outcomes tool to support goal-oriented care: a qualitative study. BMC Med Inform Decis Mak. 2021 Dec 29;21(1):366. doi: 10.1186/s12911-021-01734-0. PMID 34965860
- [Derived] Tahsin F, Tracy S, Chau E, Harvey S, Loganathan M, McKinstry B, Mercer SW, Nie J, Ramsay T, Thavorn K, Palen T, Sritharan J, Steele Gray C. Exploring the relationship between the usability of a goal-oriented mobile health application and non-usage attrition in patients with multimorbidity: A blended data analysis approach. Digit Health. 2021 Oct 5;7:20552076211045579. doi: 10.1177/20552076211045579. eCollection 2021 Jan-Dec. PMID 34868614
- [Derived] Steele Gray C, Chau E, Tahsin F, Harvey S, Loganathan M, McKinstry B, Mercer SW, Nie JX, Palen TE, Ramsay T, Thavorn K, Upshur R, Wodchis WP. Assessing the Implementation and Effectiveness of the Electronic Patient-Reported Outcome Tool for Older Adults With Complex Care Needs: Mixed Methods Study. J Med Internet Res. 2021 Dec 2;23(12):e29071. doi: 10.2196/29071. PMID 34860675
- See also: ePRO Published Protocol DOI: 10.2196/resprot.5756 (PMID: 27341765) — http://www.researchprotocols.org/2016/2/e126/